CLINICAL TRIAL: NCT01224340
Title: Active and Passive Distraction in Children Undergoing Wound Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sahlgrenska Hospital
Record Dates: First submitted 2010-10-13; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2007-05

CONDITIONS: Minor Trauma

ARMS (3):
- lollipop (Experimental): The lollipops varied in color and each color had its own flavor. The children chose between blue, green, red, orange or yellow lollipop colors. The children started to taste the lollipops approximately three to five minutes before the wound care and continued to do so during the whole session.
  Interventions: Behavioral: lollipop
- serious games (Experimental): The serious game chosen, Tux Racer, contented a penguin that collected fishes at the same time as it did slalom in a path. The player got points for collected fishes but also credits for time of flying and speed.
  Interventions: Behavioral: serious games
- control (Experimental): The participants in the control group were offered standard care without any specific distraction techniques, except consolation by the acting staff.
  Interventions: Other: control

INTERVENTIONS:
Behavioral: lollipop — The lollipops varied in color and each color had its own flavor. The children chose between blue, green, red, orange or yellow lollipop colors. The children started to taste the lollipops approximately three to five minutes before the wound care and continued to do so during the whole session.
  Arms: lollipop
Behavioral: serious games — The serious game chosen, Tux Racer, contented a penguin that collected fishes at the same time as it did slalom in a path.
  Arms: serious games
Other: control — The participants in the control group were offered standard care without any specific distraction techniques, except consolation by the acting staff.
  Arms: control

SUMMARY:
The hypothesis was that an active distraction is more effective than a passive distraction in conjunction with procedural pain in children. The specific aim in this study was to test how an active distraction, serious gaming and a passive distraction, the use of lollipops influence pain, distress and anxiety in children during wound care.

ELIGIBILITY:
Inclusion Criteria:

Children aged five to twelve were recruited from the pediatric day care unit at the Queen Silvia Children's hospital, Gothenburg, Sweden. Included children had wounds that differed in size and location but were too extensive to be handled in a primary care setting. The wound dressing procedures were standardized and the pain experiences were expected to be similar in all included children.

Exclusion Criteria:

Children with longstanding wounds, care-related pressure wounds, and wounds in body areas with decreased sensitivity were excluded from this study.Children with cognitive impairments were excluded from the study, as were children or parents who did not have a good command of Swedish.

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Self-reported pain intensity is measured on a Coloured Analogue Scale | Primary outcome, i.e. pain intensity during the wound dressing, is recorded after one wound dressing, an average time on 20 minutes.
  Primary outcome and calculation of sample size is based on self-reported pain scores. Data will be collected in conjunction with the children's first visit to the specialized wound care nurse after the trauma. Pain intensity as primary outcome is recorded at one occasion; pain intensity during the procedure is recorded after the wound care.

CONTACTS AND LOCATIONS:
Locations (1):
- The Queen Silvia Children's Hospital, Sahlgrenska University Hospital, Gothenburg, Sweden